CLINICAL TRIAL: NCT05802589
Title: Comparison of the Efficiency of Pericapsular Nerve Group Block and Unilateral Lumbar Erector Spina Plan Block Used for Postoperative Analgesia in Elective Hip Surgery: A Prospective Randomized Feasibility Study
Brief Title: Comparison of the Efficiency of PENG Block and ESP Block Used for Postoperative Analgesia in Elective Hip Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Onur Kucuk, Department of anesthesiology and reanimation, Research Assistant, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TÜTF-BAEK 2021/225
Record Dates: First submitted 2023-03-25; First posted 2023-04-06 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Pain, Postoperative; Anesthesia, Regional; Hip Surgery; Ultrasound-Guided
Keywords: Hip Surgery; Pericapsular Nerve Group Block; Lumbar Erector Spinae Plane Block; Regional Anesthesia; Ultrasound-Guided
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized, double-blind, prospective efficacy study.
Who Masked: Participant
Masking Description: Before surgery, patients were given a random number and all data were collected using this number. Group assignments were determined using simple randomization using the closed envelope technique. All data were collected blindly. The blocks were performed by the authors who did not play any role in data collection or analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (no peripheral block applied) (Active Comparator): No peripheral block was applied to this group and it was accepted as the control group. Standard multimodal analgesia and rescue analgesia according to NRS score were applied to each group.
  Interventions: Procedure: no peripheral block
- Lumbar Erector Spinae Plane Block (L-ESPB) Group (Active Comparator): Lumbar erector spinae plane block was applied to this group under ultrasound guidance. Standard multimodal analgesia and rescue analgesia according to NRS score were applied to each group.
  Interventions: Procedure: Lumbar Erector Spinae Plane Block
- Pericapsular Nerve Group Block (PENGB) Group (Active Comparator): Pericapsular nerve group block was applied to this group under ultrasound guidance. Standard multimodal analgesia and rescue analgesia according to NRS score were applied to each group.
  Interventions: Procedure: Pericapsular Nerve Group Block

INTERVENTIONS:
Procedure: Lumbar Erector Spinae Plane Block — Erector spinae plane block was applied with a 22G/80 mm block needle (Stimuplex A, Braun, Melsungen, Germany) using in-plane technique using a convex USG transducer from the 4th lumbar vertebral level.
  Arms: Lumbar Erector Spinae Plane Block (L-ESPB) Group
Procedure: Pericapsular Nerve Group Block — Pericapsular nerve group block was performed using a 22G/80 mm block needle (Stimuplex A, Braun, Melsungen, Germany) and a convex USG transducer using an in-plane technique under the iliopsoas muscle in the plane between the iliopsoas tendon and the periosteum and between the anterior inferior iliac spine and the iliopubic eminence.
  Arms: Pericapsular Nerve Group Block (PENGB) Group
Procedure: no peripheral block — No peripheral block was applied. Standard multimodal analgesia method was applied.
  Arms: Control Group (no peripheral block applied)

SUMMARY:
The aim of the study is to determine whether the traditional intravenous analgesia technique or the ultrasound-guided pericapsular nerve group block or the unilateral erector spina plane block technique is superior in postoperative analgesia management in the hip operation procedure that requires preoperative and postoperative severe analgesia. In this way, by preventing the health problems that may occur due to the pain of the patients after the operation; to provide benefits for the early mobilization of patients, shortening the hospital stay, reducing the cost and increasing patient satisfaction.

DETAILED DESCRIPTION:
Hip arthroplasty (HA) is one of the most successful orthopedic procedures applied today to improve the patient's functional status and quality of life. In patients with hip pain due to various conditions, HA can relieve pain, restore function, and improve quality of life. In the USA alone, approximately 500,000 HA is performed each year. With the increase in the elderly population, HA surgeries have also increased, but despite the developing methods, a gold standard has not been determined for anesthesia and analgesia methods. Appropriate pain management for surgical patients contributes to early mobilization, shortened hospital stay, reduced cost and increased patient satisfaction, while inadequate treatment of pain has detrimental short- or long-term health effects. Therefore, minimizing postoperative pain has become more important for healthcare providers in recent years. Therefore, postoperative pain control can be achieved with balanced and effective analgesia. For this purpose, various analgesia techniques have been used to prevent postoperative pain. The superiority of the techniques to each other varies according to the type of surgery and the combination of techniques applied. Opioids, which are the most widely used to prevent inadequate pain treatment leading to various comorbidities, cause pharmacodynamic results due to physiological changes and serious side effects due to concomitant diseases in patients. In recent years, peripheral nerve blocks have been used in the management of postoperative pain in hip surgeries. Erector spina plane block and pericapsular nerve group block are the most reliable and proven blocks used in hip operations.

The aim of the study is to determine whether traditional intravenous analgesia technique, ultrasound-guided pericapsular nerve group block or unilateral erector spina plane block technique is superior in postoperative analgesia management in hip operation procedure requiring preoperative and postoperative severe analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective hip or proximal femoral surgery
* 18-89 years old
* Patients with the American Society of Anesthesiology physical condition classification score (ASA) I-III

Exclusion Criteria:

* Patients who do not agree to consent
* Patients who requested to be excluded from the study
* Patients allergic to local anesthetics
* Those with infection at the intervention site
* Those who weigh <30 kg
* Those aged <18 years
* Those with an ASA physical condition of 4 or higher
* People with dementia or cognitive impairment
* Patients with bleeding diathesis pathology
* Patients using chronic opioids or corticosteroids
* Patients whose surgical procedure takes <60 minutes or >180 minutes

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | postoperative 24 hours score change
  NRS was used to assess postoperative pain. The NRS is a segmented numerical version of the visual analog scale (VAS), in which the respondent chooses an integer (0-10 integer) that best reflects the intensity of his pain. It is considered a one-dimensional measure of pain intensity in adults. It is an 11-point numerical scale. It ranges from "0" representing no pain to "10" representing extreme pain.

SECONDARY OUTCOMES:
Additional Analgesia | postoperative 24 hours additional analgesic drug administration
  Analgesic drugs administered in the first 24 hours in addition to the routine multimodal analgesia procedure were recorded.
5-point likert satisfaction scale | postoperative 24th hour
  The patient's satisfaction with postoperative pain treatment will be recorded. 5 options; very dissatisfied, dissatisfied, neither dissatisfied or satisfied, satisfied, very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: ONUR KÜÇÜK, specialist, Principal Investigator — Trakya University
Locations (1):
- Trakya University, Edirne, Centrum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No